CLINICAL TRIAL: NCT04701424
Title: An Open-label, Single-centre, Randomised, 2-period Cross-over Study to Assess the Efficacy, Safety and Utility of Fully Closed-loop Insulin Delivery in Comparison With Standard Care in Adults With Type 2 Diabetes Not Requiring Dialysis
Brief Title: Closed-loop in Adults With T2D Not Requiring Dialysis
Acronym: AP-Renal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Dr Roman Hovorka, Professor of Metabolic Technology, University of Cambridge
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RG97920
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; type 2 diabetes; closed-loop; artificial pancreas; insulin pump therapy; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Closed loop insulin delivery (Experimental): Unsupervised home use of day and night fully automated closed loop insulin delivery system (CamAPS HX) for 8 weeks
  The CamAPS HX closed-loop system comprises:
  Dana insulin pump (Diabecare, Sooil, Seoul, South Korea) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA) An Android smartphone hosting CamAPS HX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump Glooko/Diasend cloud upload system to monitor CGM/insulin data
  Interventions: Device: CamAPS HX Closed-loop
- Standard therapy (Active Comparator): Participants in the control arm will continue to follow their current diabetes management plan for the 8 week study period. Participants will be wear a masked continuous glucose monitoring (CGM) system during the 8 week study period
  Interventions: Other: Multiple Daily Insulin Injections (Control)

INTERVENTIONS:
Device: CamAPS HX Closed-loop — The CamAPS HX closed-loop system comprises:
  Dana insulin pump (Diabecare, Sooil, Seoul, South Korea) Dexcom G6 real-time CGM sensor (Dexcom, Northridge, CA, USA) An Android smartphone hosting CamAPS HX Application with the Cambridge model predictive control algorithm and communicating wirelessly with the insulin pump Glooko/Diasend cloud upload system to monitor CGM/insulin data.
  Arms: Closed loop insulin delivery
Other: Multiple Daily Insulin Injections (Control) — Multiple Daily Insulin Injections with masked Dexcom G6 CGM sensor (Dexcom, Northridge, CA, USA)
  Arms: Standard therapy

SUMMARY:
The main objective of this study is to determine the efficacy, safety and utility of fully automated closed-loop glucose control in the home setting over an 8 week period in adults with type 2 diabetes (T2D). This study builds on previous and on-going studies of closed-loop systems that have been performed in Cambridge in adults with type 1 diabetes in the home setting, and in adults with type 2 diabetes in the inpatient setting.

This is an open-label, single centre, randomised, cross-over study, involving two home study periods during which glucose levels will be controlled either by a fully automated closed-loop system or by participants' usual insulin therapy in random order. Each treatment arm is 8 weeks long with a 2-4 week washout period between treatments. A total of up to 30 participants with T2D will be recruited through outpatient clinics to allow for 24 completed participants available for assessment.

Participants will receive appropriate training by the research team on the safe use of the study devices (insulin pump and continuous glucose monitoring (CGM) and closed-loop insulin delivery system). Participants in the control arm will continue with standard therapy and will wear a blinded CGM system.

The primary outcome is time spent with glucose levels in the target range between 3.9 and 10.0 mmol/L as recorded by CGM. Secondary outcomes are the time spent with glucose levels above and below target, as recorded by CGM, and other CGM-based metrics in addition to insulin requirements. Safety evaluation comprises the tabulation of severe hypoglycaemic episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or over
2. Diagnosis of type 2 diabetes using standard diagnostic practice
3. Current treatment with subcutaneous insulin
4. Screening HbA1c ≤ 11% (97mmol/mol) on analysis from local laboratory
5. Subject is willing to perform regular finger-prick blood glucose monitoring
6. Willingness to wear study devices
7. Literate in English

Exclusion Criteria:

1. Physical or psychological condition likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator
2. Known or suspected allergy to insulin
3. Lack of reliable telephone facility for contact
4. Pregnancy, planned pregnancy, or breast feeding
5. Severe visual impairment
6. Severe hearing impairment
7. Medically documented allergy towards the adhesive (glue) of plasters
8. Serious skin diseases located at places of the body, which potentially are possible to be used for localisation of the glucose sensor
9. Illicit drugs abuse
10. Prescription drugs abuse
11. Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Time in the target glucose range (3.9 to 10.0 mmol/l) | 8 week intervention period
  Percentage of time spent with sensor glucose readings in the target range from 3.9 to 10.0mmol/l

SECONDARY OUTCOMES:
Time spent above target glucose (10.0 mmol/l) | 8 week intervention period, both arms
  Percentage of time spent with sensor glucose readings above target glucose (10.0 mmol/l)
Mean glucose | 8 week intervention period, both arms
  Mean sensor glucose level
Time spent in hypoglycaemia (<3.9 mmol/l) | 8 week intervention period, both arms
  Percentage of time spent with sensor glucose readings <3.9 mmol/L
Standard deviation of glucose levels | 8 week intervention period, both arms
  Standard deviation of glucose levels
Coefficient of variation of glucose levels | 8 week intervention period, both arms
  Coefficient of variation of glucose levels
Time spent below <3.0 mmol/l | 8 week intervention period, both arms
  Percentage of time spent with sensor glucose readings <3.0 mmol/l
Time in hyperglycaemia > 16.7 mmol/l | 8 week intervention period, both arms
  Percentage of time with glucose levels in hyperglycaemia > 16.7 mmol/l
Time in significant hyperglycaemia (> 20 mmol/l) | 8 week intervention period, both arms
  Percentage of time with glucose levels in significant hyperglycaemia (> 20 mmol/l)
Glycated haemoglobin (HbA1c) | 8 week intervention period, both arms
  HbA1c measured at the end of each study period
Total insulin dose | 8 week intervention period, both arms
  Average daily total insulin requirements

OTHER OUTCOMES:
Number of episodes of severe hypoglycaemia | 8 week intervention period, both arms
  Safety evaluation
Number of subjects experiencing severe hypoglycaemia | 8 week intervention period, both arms
  Safety evaluation
Frequency and nature of other adverse events or serious adverse events | 8 week intervention period, both arms
  Safety evaluation
Percentage of time of closed-loop operation | 8 week intervention period, both arms
  Utility evaluation
Percentage of time of CGM availability | 8 week intervention period, both arms
  Utility evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Roman Hovorka, PhD, Principal Investigator — University of Cambridge
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised data may be shared with third parties (EU or non-EU based) for the purposes of advancing management and treatment of diabetes.

REFERENCES:
- [Derived] Daly AB, Boughton CK, Nwokolo M, Hartnell S, Wilinska ME, Cezar A, Evans ML, Hovorka R. Fully automated closed-loop insulin delivery in adults with type 2 diabetes: an open-label, single-center, randomized crossover trial. Nat Med. 2023 Jan;29(1):203-208. doi: 10.1038/s41591-022-02144-z. Epub 2023 Jan 11. PMID 36631592